CLINICAL TRIAL: NCT06317415
Title: Effect of Health Education on Non-prescription Antibiotic Use Among the Public: a Cluster Randomized Controlled Trial
Brief Title: Intervention on Non-prescription Antibiotic Use Among the Public
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: Fuyong People's Hospital, Bao 'an District, Shenzhen City, Guangdong (Unknown)
Responsible Party: Principal Investigator, Xiaoxv Yin, PhD, Professor, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: HuazhongU20240312
Record Dates: First submitted 2024-03-12; First posted 2024-03-19 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Non-Prescription Drug Misuse; Antibiotic Use
Keywords: Cluster randomized trial; Non-prescription; antibiotic
MeSH Terms: conditions — Drug Misuse

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Behavioral: WeChat-based health education on antibiotic use
- control group (Placebo Comparator)
  Interventions: Behavioral: Regular public health education

INTERVENTIONS:
Behavioral: WeChat-based health education on antibiotic use — Health education based on the WeChat platform includes popular science articles on WeChat public Platform and health education videos.
  Arms: Intervention group
Behavioral: Regular public health education — Health education information on the prevention and control of common chronic diseases
  Arms: control group

SUMMARY:
The purpose of this study is to test the effectiveness of health education int led by community health workers for non-prescription antibiotic use among the public. In this two arm cluster randomised trial, In this two-arm cluster randomized controlled trial, 22 communities were randomly allocated in a 1:1 ratio to intervention and control groups. In the intervention group, family doctors will conduct WeChat-based health education on responsible use of antibiotic for the participants. In the control group, only routine public health education will be provided without any involvement in antibiotic use. The primary outcome is the incidence of antibiotic use without prescription in the past month.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 75 years old;
* Local residents (residing for more than 6 months) with no plans for employment, study, or relocation in the next six months;
* Having normal cognitive, comprehension, and independent communication abilities, and voluntarily participating in this study;
* Able to use WeChat independently or with guidance from family members.

Exclusion Criteria:

* Unable to comprehend the purpose of the survey, unwilling to cooperate, or lacking willingness to provide honest answers to questions;
* Illiterate, severely physically disabled, or lacking necessary comprehension abilities;
* Healthcare professionals, such as doctors, nurses, pharmacists, etc.;
* Individuals with autoimmune diseases or hereditary diseases affecting the use of common medications;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1550 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Rate of non-prescription antibiotic use among the public | within one month
  Rate of Antibiotic use without prescription in the past month measured by self-designed questionnaire。

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoxv Yin, Principal Investigator — Huazhong University of Science and Technology
Locations (1):
- Fuyong People's Hospital, Shenzhen, Guangdong, China